CLINICAL TRIAL: NCT01037530
Title: A Double Blind, Randomised, Placebo Controlled Trial to Study the Clinical and Cost Effectiveness of the Angiotensin Converting Enzyme Inhibitor, Ramipril, in Intermittent Claudicants
Brief Title: Clinical and Cost Effectiveness of ACE Inhibitor, Ramipril, in Intermittent Claudicants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05102009; 2009-016600-23 (Registry Identifier: European Clinical Trials Database (EudraCT))
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2022-04

CONDITIONS: Intermittent Claudicants
Keywords: ACE inhibitors; Intermittent claudication; Ramipril
MeSH Terms: conditions — Intermittent Claudication | interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramipril (Experimental)
  Interventions: Drug: Ramipril
- Placebo (Placebo Comparator)
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — 5 mg/day for 2 weeks then 10 mg/day for 22 weeks

SUMMARY:
The investigators are conducting a randomised controlled trial to investigate the clinical and cost effectiveness of Ramipril which is an anti-hypertensive medication in patients with intermittent claudication. The investigators aim to recruit 78 participants in total. The investigators will randomise the 78 participants into two groups: Ramipril group with 39 participants and Placebo group with 39 participants. The investigators will measure Ramipril's effect on walking by doing a simple treadmill test and measuring the maximum walking distance the participant can walk. The investigators also want to examine Ramipril's effect on arterial function, cardiovascular prognosis, quality of life and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral intermittent leg claudication which was stable for the last 6 months.
* Patients with ABPI < 0.9 at rest at least in one leg.
* BP ≤ 160/90 and a stable medication regimen for the last 6 months.
* Able to give informed consent
* Able to comply with study protocol

Exclusion Criteria:

* Documented bilateral renal artery stenosis
* Unlikely to be compliant with medication or follow up as determined by the recruiting institution.
* Pregnancy
* Patients with critical limb ischemia (This includes patients with ischaemic rest pain and ulceration > 2 weeks and/or a resting ankle pressure < 50mmHg- Grades II and III according to Rutherford et al 1997.[56].
* Patients who had a recent (less than 3 months) angioplasty or bypass surgery
* Patients who are unable to perform a treadmill test due to a limiting heart, respiratory or arthritic disease
* History of angioneurotic oedema
* Currently taking ACE inhibitor or Angiotensin receptor blocker
* Contraindication to ACE inhibitor
* History of ACE inhibitor intolerance
* A creatinine rise of > 30% from baseline and/or Potassium > 5.9 mmol/l
* Unwillingness to participate.
* Level 1 evidence for ACE inhibitor treatment, including:
* Documented heart failure, left ventricular dysfunction or ejection fraction <35% on previous echocardiography

  * Uncontrolled hypertension, BP > 160mmHg systolic or 100mmHg diastolic on 3 separate readings measured after 10 minutes rest on 2 separate occasions
  * Recent (< 3months) myocardial infarction or stroke
  * Chronic renal impairment (serum creatinine > 250 micromol/l)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Chetter, MD, FRCS, Principal Investigator — University of Hull
Locations (1):
- Hull and East Yorkshire Hospitals, Hull, Yorkshire, United Kingdom

REFERENCES:
- [Result] Shahin Y, Cockcroft JR, Chetter IC. Randomized clinical trial of angiotensin-converting enzyme inhibitor, ramipril, in patients with intermittent claudication. Br J Surg. 2013 Aug;100(9):1154-63. doi: 10.1002/bjs.9198. PMID 23842829
- See also: Related publications — http://www.ncbi.nlm.nih.gov/pubmed/21195215

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ramipril | Placebo
Started | 14 | 19
Completed | 12 | 17
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramipril | Placebo | Total
Number analyzed (Participants) | 14 | 19 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (8.2) | 64.7 (7.7) | 64.55 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Walking Distance (MWD).
Description: The primary outcome measure for this trial is the Maximum Walking Distance (MWD). Treadmill exercise test will be used to estimate the maximum distance the participant can walk at a speed of 2.5 km/h with a 10
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Metres
Arm/Group | Ramipril | Placebo
Number analyzed (Participants) | 14 | 19
Metres | 137 [110 to 213] | 143 [72 to 213]

2. Secondary Outcome: Other Clinical Indicators of Lower Limb Ischaemia: a) Patient Reported Walking Distance (PRWD) b) Treadmill Intermittent Claudication Distance (ICD) c) Ankle Brachial Pressure Index at Rest (ABPI- r) and Following Treadmill Testing (ABPI - t)
Time Frame: Baseline
Reporting Status: Not Posted

3. Secondary Outcome: Quality of Life: a) Generic - Measured Using the SF36, SF8 and EuroQol (EQ5D) Instruments b) Disease Specific - Measured Using the VascuQol
Time Frame: 0,2,6,24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Cardiovascular Prognosis Using: a) Framingham, PROCAM, QRISK and Manchester Charts Scoring Systems b) B-type Natriuretic Peptide (BNP) and N- Terminal Prohormone BNP (NT-proBNP) and a Lipid Profile ( LDL, HDL, Total Cholesterol, Triglycerides)
Time Frame: 0,2,6,24 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Markers of Endothelial Function and Ischaemia Reperfusion a) IL6 b) Soluble Intercellular Adhesion Molecule-1 (sICAM -1) c) sE Selectin d) Urine Albumin Creatinine Ratio ( UACR)
Time Frame: 0,2,6,24 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Arterial Effects: a) Arterial Stiffness by Measuring the Pulse Wave Velocity and Assessing the Effects on the Extracellular Matrix by Measuring Metalloproteinases (MMPs) and Tissue Inhibitor Metalloproteinases (TIMPs). b) Flow Mediated Vasodilatation
Time Frame: 0,2,6,24 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Health Economics (Cost Effectiveness / Utility)
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ramipril | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/19
Other Adverse Events (participants affected / at risk) | 6/14 | 0/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramipril (N=14) | Placebo (N=19)
Cough (Cardiac disorders) | 4 (4) | 0 (0)
Dizziness (General disorders) | 1 (1) | NA
Hyperkalaemia (Endocrine disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes